CLINICAL TRIAL: NCT00002646
Title: PHASE III DOUBLE-BLIND, PLACEBO-CONTROLLED, PROSPECTIVE RANDOMIZED COMPARISON OF ADJUVANT THERAPY WITH TAMOXIFEN VS. TAMOXIFEN AND FENRETINIDE IN POSTMENOPAUSAL WOMEN WITH INVOLVED AXILLARY LYMPH NODES AND POSITIVE RECEPTORS
Brief Title: Hormone Therapy in Treating Postmenopausal Women With Receptor-Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network); North Central Cancer Treatment Group (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064156; E-EB193; CLB-9443; NCCTG-953052; SWOG-9514; INT-0151
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2010-10

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fenretinide; Tamoxifen

INTERVENTIONS:
Drug: fenretinide
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen. Combining chemotherapy with hormone therapy may kill more tumor cells. Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of fenretinide may be an effective way to prevent the recurrence of breast cancer. It is not yet known whether tamoxifen plus fenretinide is more effective than tamoxifen alone for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of tamoxifen plus fenretinide with tamoxifen alone in treating postmenopausal women who have stage II or stage III breast cancer that is estrogen receptor positive and/or progesterone receptor positive.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare disease free survival and overall survival of postmenopausal women with stage II or IIIA breast cancer treated with tamoxifen (TMX) and fenretinide (HPR) vs TMX and placebo. II. Gain wider experience in the use and toxicity of combined TMX/HPR in these patients. III. Obtain tumor tissue samples, as feasible, from these patients for future biologic studies.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified by participating institution, age (under 70 vs 70 and over), node dissection (yes vs no), number of involved nodes (0 vs 1-3 vs 4 or more), and number of removed nodes (1-5 vs 6 or more). All patients receive oral tamoxifen daily for at least 5 years, beginning immediately after randomization. Patients also receive either oral fenretinide or oral placebo daily for 5 years, beginning within 2 weeks after completion of any radiotherapy, or within 2 weeks of randomization, if no radiation. Patients are followed during and after treatment every 4 months for 2 years, every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 1,500 patients will be accrued for this study over approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the breast Pathologic stage T1-3, N1-2, M0 No clinical or pathologic T4 disease No primary tumor fixed to chest wall No axillary nodes fixed to chest wall or neurovascular bundle No preoperative arm edema No clinical skin involvement (microscopic focal dermal invasion or dermal lymphatic involvement eligible) No clinical N2 disease Modified radical mastectomy or lumpectomy required prior to entry Sentinel node biopsy allowed Randomization required within 12 weeks from definitive surgery Surgery dated from mastectomy or axillary dissection for lumpectomy No positive deep mastectomy margins Radiotherapy planned within 12 weeks following axillary node dissection for lumpectomy patients Synchronous bilateral breast cancer eligible If tumor is at least 2 cm, then nodes not involved If no tumor is at least 2 cm, then at least 1 node must be involved Both invasive primaries receptor-positive Previously treated, noninvasive breast cancer eligible No prior invasive breast cancer No adenoid cystic, squamous, or sarcomatous histology Hormone receptor status: Estrogen- or progesterone-receptor positive, i.e.: At least 10 fmole/mg cytosol protein by ligand-binding assay OR Receptor positive by immunocytochemistry

PATIENT CHARACTERISTICS: Age: 65 and over OR Postmenopausal and ineligible/inappropriate for or declined other active node positive adjuvant studies Sex: Female Menopausal status: Postmenopausal, defined as: At least 1 year since last menstrual period Hysterectomized with bilateral oophorectomy Hysterectomized with 1 or both ovaries remaining and either: Over 60 FSH in postmenopausal range Not surgically castrated, under 60, and on HRT FSH elevated 2 weeks after HRT discontinued Performance status: Not specified Life expectancy: At least 7 years except for breast cancer Hematopoietic: WBC greater than 3,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL AST less than 2 times normal Renal: Creatinine no greater than 2.0 mg/dL BUN no greater than 25.0 mg/dL Other: No extensive macular degeneration on exam within 1 year of entry, e.g.: No exudative or atrophic macular lesions that reduce corrected vision to less than 20/40 Health adequate for protocol treatment No nutritional supplementation except single daily multivitamin No other vitamin A supplements Gynecologic exam within the past year required of women who retain a uterus No second malignancy within the past 10 years except: Inactive nonmelanomatous skin cancer Carcinoma in situ of the cervix Prior noninvasive contralateral breast cancer

PRIOR CONCURRENT THERAPY: No prior chemotherapy or hormonal therapy for breast cancer except: Up to 1 month of tamoxifen if started by a non participating physician At least 2 weeks since hormone replacement therapy No concurrent megestrol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 1995-10; Primary Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melody A. Cobleigh, MD, Study Chair — Rush University Medical Center; George Thomas Budd, MD, Study Chair — The Cleveland Clinic; Mark L. Graham, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center; James N. Ingle, MD, Study Chair — Mayo Clinic
Locations (85):
- United States (85):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Rao RD, Cobleigh MA, Gray R, Graham ML 2nd, Norton L, Martino S, Budd GT, Ingle JN, Wood WC. Phase III double-blind, placebo-controlled, prospective randomized trial of adjuvant tamoxifen vs. tamoxifen and fenretinide in postmenopausal women with positive receptors (EB193): an intergroup trial coordinated by the Eastern Cooperative Oncology Group. Med Oncol. 2011 Dec;28 Suppl 1(Suppl 1):S39-47. doi: 10.1007/s12032-010-9682-1. Epub 2010 Sep 28. PMID 20878269
- [Result] Cobleigh MA, Gray R, Graham M, et al.: Fenretinide (FEN) vs placebo in postmenopausal breast cancer patients receiving adjuvant tamoxifen (TAM), an Eastern Cooperative Oncology Group Phase III Intergroup Trial (EB193, INT-0151). [Abstract] Proceedings of the American Society of Clinical Oncology 19: A328, 2000.